CLINICAL TRIAL: NCT06109688
Title: Effect of Lactoferrin Supplementation on Urinary Tract Infections in Infants: a Randomised, Double-blind, Placebo-controlled Trial.
Brief Title: Effect of Lactoferrin Supplementation on Urinary Tract Infections in Infants.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Collaborators: Pharmabest Sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0254/297/2014
Record Dates: First submitted 2020-04-27; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Urinary Tract Infections in Children
Keywords: urinary tract infections; infants; lactoferrin
MeSH Terms: conditions — Urinary Tract Infections | interventions — Lactoferrin; maltodextrin

STUDY DESIGN:
Intervention Model Description: patients with Urinary Tract Infections were recruited subjects were randomized into two groups:
  * the experimental group received bLF
  * the control group received placebo without bLF
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bovine lactoferrin (Experimental): Sachets with bovine lactoferrin at a dosage of 100 mg/day for a period of 4 weeks.
  Interventions: Dietary Supplement: Bovine Lactoferrin
- Placebo (Placebo Comparator): Matched sachets with maltodextrin for a period of 4 weeks.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Bovine Lactoferrin — Orally intake 1 sachet per day for 4 weeks. Lactoferrin will be dissolved in human milk or infant formula or in a 5% glucose solution.
  Other Names: Lactoferrin 100 mg
  Arms: Bovine lactoferrin
Dietary Supplement: placebo — Orally intake 1 sachet per day for 4 weeks. Maltodextrin will be dissolved in human milk or infant formula or in a 5% glucose solution.
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
The aim of the study was to evaluate the efficacy of orally administered bovine lactoferrin (bLF) on Urinary Tract Infections in neonates and infants. Fifty-five patients with urinary tract infection were randomized to receive either bLF (n = 27) or an identical placebo (n = 28) for 4 weeks. The patients were assessed clinically and laboratory.

DETAILED DESCRIPTION:
This study was a prospective randomized controlled trial at a single university medical center. Participants were neonates or infants with Urinary Tract Infection (UTI) admitted to the Neonatal and Infant Pathology Department of Children's University Hospital in the period from July 2015 to December 2017. The intervention was bovine lactoferrin at a dosage of 100 mg/day for a period of 4 weeks compared with placebo in a control group.

During hospital treatment, laboratory tests were performed to evaluate the activity of inflammatory markers (C-reactive protein, procalcitonin, Interleukin-6 and Interleukin-8 levels and white blood cell count).

Fifty-five patients heve been included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infants with symptoms of Urinary Tract Infection.
* Active infection at enrollment, confirmed and documented in medical record.
* Children with Urinary Tract Infection treated according to current recommendations.

Exclusion Criteria:

* Unconfirmed Urinary Tract Infection.
* Critical illness and/or hemodynamic instability.
* Allergy or sensitivity to lactoferrin or bovine derived proteins or bovine milk.
* Children whose parents/guardians decline to participate.

Ages: 7 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Monitoring of parameters of inflammation. | at baseline, after 5 days of treatment
  C-reactive protein and procalcitonin levels in both groups. Comparing possible change.
Influence of lactoferrin on Interleukin-6 and Interleukin-8. | at baseline, after 5 days of treatment
  Levels of Interleukin in both groups. Comparing possible change.
Effect of lactoferrin on white blood cells. | at baseline, after 5 days of treatment
  To assess the change in the number of leukocytes, neutrophils, lymphocytes, monocytes, eosinophils and basophils.
Effect of lactoferrin on urinary inflammatory markers. | at baseline, after 5 days of treatment
  The presence of bacteria in urine and semi-quantitative measurement of white blood cells count in urine.

SECONDARY OUTCOMES:
To evaluate the efficacy of lactoferrin in the reduction of probable recurrence of Urinary Tract Infection. | 1 month
  The number of recurrent Urinary Tract Infections occur due to bacterial reinfection or bacterial persistence.
The number of days of hospitalization. | 1 month
  Length of stay. Comparing possible differences in groups.
Evaluation of the safety of the administration of lactoferrin by monitoring possible adverse effects. | 1 month
  Incidence, frequency and severity of treatment emergent adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Kuźma, Principal Investigator — Department of Neonate and Infant Pathology, Medical University of Lublin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manzoni P, Dall'Agnola A, Tome D, Kaufman DA, Tavella E, Pieretto M, Messina A, De Luca D, Bellaiche M, Mosca A, Piloquet H, Simeoni U, Picaud JC, Del Vecchio A. Role of Lactoferrin in Neonates and Infants: An Update. Am J Perinatol. 2018 May;35(6):561-565. doi: 10.1055/s-0038-1639359. Epub 2018 Apr 25. PMID 29694997
- [Background] Artym J, Zimecki M. [The role of lactoferrin in the proper development of newborns]. Postepy Hig Med Dosw (Online). 2005;59:421-32. Polish. PMID 16106243
- [Background] Balighian E, Burke M. Urinary Tract Infections in Children. Pediatr Rev. 2018 Jan;39(1):3-12. doi: 10.1542/pir.2017-0007. No abstract available. PMID 29292282
- [Background] Garout WA, Kurdi HS, Shilli AH, Kari JA. Urinary tract infection in children younger than 5 years. Etiology and associated urological anomalies. Saudi Med J. 2015 Apr;36(4):497-501. doi: 10.15537/smj.2015.4.10770. PMID 25828291
- [Background] Renata Y, Jassar H, Katz R, Hochberg A, Nir RR, Klein-Kremer A. Urinary concentration of cytokines in children with acute pyelonephritis. Eur J Pediatr. 2013 Jun;172(6):769-74. doi: 10.1007/s00431-012-1914-2. Epub 2013 Feb 7. PMID 23389820
- [Background] Krzemien G, Szmigielska A, Turczyn A, Panczyk-Tomaszewska M. Urine interleukin-6, interleukin-8 and transforming growth factor beta1 in infants with urinary tract infection and asymptomatic bacteriuria. Cent Eur J Immunol. 2016;41(3):260-267. doi: 10.5114/ceji.2016.63125. Epub 2016 Oct 25. PMID 27833443
- [Background] Miguel-Bayarri V, Casanoves-Laparra EB, Pallas-Beneyto L, Sancho-Chinesta S, Martin-Osorio LF, Tormo-Calandin C, Bautista-Rentero D. Prognostic value of the biomarkers procalcitonin, interleukin-6 and C-reactive protein in severe sepsis. Med Intensiva. 2012 Nov;36(8):556-62. doi: 10.1016/j.medin.2012.01.014. Epub 2012 Apr 10. English, Spanish. PMID 22495097